CLINICAL TRIAL: NCT01576159
Title: The Effect of Mechanical Loading During Sports Exercises on Degradation of Human Articular Cartilage
Brief Title: Serum Cartilage Oligomeric Matrix Protein Levels After 12 Weeks of Different Exercises
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Middle East Technical University (Other)
Responsible Party: Principal Investigator, Feza Korkusuz, Prof. Dr., Middle East Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BAPK06K07K03K00K17; 107S112 (Other: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2012-04-09; First posted 2012-04-12 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis; Articular Cartilage Disorder of Knee; Degenerative Lesion of Articular Cartilage of Knee
Keywords: Biochemical Marker; Fitness Exercises; Impact; Articular Cartilage
MeSH Terms: conditions — Osteoarthritis; Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High-Impact Loading (Experimental): Performed high-impact running exercise during intervention period.
  Interventions: Other: Running exercise
- Moderate-Impact Loading (Experimental): Performed moderate-impact cycling exercise during intervention period.
  Interventions: Other: Cycling exercise
- Non-Impact Loading (Experimental): Performed low-impact swimming exercise during intervention period.
  Interventions: Other: Swimming Exercise
- Control Group (No Intervention): Didn't participate any organized physical exercises

INTERVENTIONS:
Other: Running exercise — During this type of exercise intervention, subjects performed weight-bearing exercise. This group participated in sessions of 40-min per day, three days per week, for a period of 12 weeks
  Arms: High-Impact Loading
Other: Cycling exercise — During this type of exercise intervention, subjects performed a partial weight-bearing exercise. This group participated in sessions of 40-min per day, three days per week, for a period of 12 weeks
  Arms: Moderate-Impact Loading
Other: Swimming Exercise — During this type of exercise intervention, subjects performed a non-weight bearing exercise. This group participated in sessions of 40-min per day, three days per week, for a period of 12 weeks
  Arms: Non-Impact Loading

SUMMARY:
Acute effects of physical exercise on the deformational behavior of articular cartilage and changes in cartilage oligomeric matrix protein (COMP) are definite. However, conclusive positive effects of fitness exercise on functional adaptation of articular cartilage have not been proved.Therefore, in this parallel-group randomized control trial, the investigators tested the hypothesis that adequate amount of physical exercise with enough impact would be able to stimulate the functional behavior of articular cartilage.

The investigators evaluated 44 healthy males for their physical fitness levels and their blood samples were obtained before, immediately after and 0.5 h after a 30-min walking exercise. Thereafter, participants were assigned to the running, the cycling, the swimming and the control groups. At the end of 12-weeks of intervention, same measurement procedures were applied. Mixed repeated-measures ANOVA design was used for statistics. (Level of evidence: 2)

DETAILED DESCRIPTION:
Design

A prospective, parallel-group randomized control trial was designed. Mustafa Kemal University (MKU) Ethical Board approved the study (B.30.2.MKU.0.01.01.00/255). The exact nature of the study was explained to participants and they were asked to sign a written consent. The tests were carried out at Middle East Technical University Medical Center, Ankara, Turkey between January and June 2008. The independent variables were groups (n=4) and time (n=2). The dependent variable was serum cartilage oligomeric matrix protein (COMP) levels measured at three phases of exercise: before (Recovery), immediately after (Fatigue), and 30-min after the exercise (Regeneration). Participants were subjected to the following tests prior to and at the end of the intervention period: body mass index (BMI), isokinetic leg muscle strength, maximum oxygen consumption (VO2max) and serum COMP levels.

Participants

115 applicants volunteered to take part in this study. Eligibility screening was performed according to inclusion criteria. From 104 eligible applicants, 48 healthy, sedentary male university students aged between 18 to 25 years old (Mage = 21.8±1.9) were selected by a simple drawing. However, study completed with 44 participants, because of 4 dropouts. Participants were randomly assigned in 1:1:1:1 ratio to parallel groups, three exercise groups (swimming, cycling and running) and one control. In order to have a random allocation, each participant received a number unknown to researchers which was written on a piece of paper and then drawn from a box that allowed to assign individuals to the control and exercise groups. Baseline blood samples were stored in -80°C and they were not analyzed during participants' allocation. Exclusion criteria, surveyed by a questionnaire, were: osteoarthritis, rheumatoid arthritis or other inflammatory joint disease, intra-articular steroid injection, mal-alignment of the knees (varus/valgus) larger than 15°, and recent (within six months) fracture of lower extremity. Active athletes and volunteers with previous sports background were not included. During the intervention period, one participant was excluded from the study because of sudden kidney disease and another one decided to withdraw from further participation. In addition, two participants were excluded from the study before biochemical analyses since one subject from running group didn't meet minimum requirement of 75% of exercise session attendance, and one subject from control group didn't complete the posttests. Descriptive data of participants are presented in.

Interventions

After the first measurements, participants were randomly and equally assigned to the swimming, the running, the cycling and the control groups. All exercise groups participated in sessions of 40-min per day, three days per week, for a period of 12 weeks. Each session began with a five minutes warm-up, continued with a main set of 30-min exercise at their individual target heart rate zone (60-70% of heart rate reserve), and finished with a five minute cool-down period. The individual target heart rate zone was determined according to the Guidelines for Exercise Testing and Prescription of American College of Sport Medicines [1]. Swimming exercises composed of front crawl swimming and kicking drills. During the main sets, the participants performed front-crawl swimming at their individual heart rate zones which were determined by the Karvonen formula [2]. Cyclers exercised between 60-80 repetition per minute (RPM) on an ergometer (Monark E 834, Varberg, Sweden), which was adjusted for each individual in order to maintain the target heart rate zone. The running group participants exercised on a treadmill with a 1.5 % incline. The speed of the treadmill was determined according to individual heart rate zone. Throughout the 12 weeks of training, Heart Rate Reserves (HRR) was held constant (60-70%) while the speed increased according to individual progression. Individuals of the control group were instructed not to participate in any organized or structured exercise during the 12 weeks of intervention.

Physical and Physiological Measurements

Body Mass Index was calculated as the ratio of body weight to height square (Heyward & Stolarczyk 1996). VO2max was measured by the standard Bruce Protocol (Bruce, Kusumi & Hosmer 1973) on a Jager LE 200 CE (Hochberg, Germany) treadmill. Measurements were performed with the VIASYS Healthcare ergospirometry line using the MasterScreen CPX (Wuerzburg, Germany) device. Results were presented in ml/kg/min (milliliters of oxygen per kilogram of body weight per minute). Isokinetic quadriceps strength was recorded with the Biodex System Dynamometer (Biodex Medical Inc, Shirley, NY). Participants were placed in a comfortable position that allowed unrestricted motion of the knee from 90 degrees of flexion to terminal extension on a bicycle ergometer, and asked to warm-up for five minutes at which point they stretched their extremities. Before the test trials, participants were instructed to perform their maximum efforts. Then five isokinetic concentric knee flexion and extension at 60°/sec with their dominant legs were recorded. After, peak torque to body weight ratio (PT/BW) was measured.

Blood Sampling and Enzyme-Linked Immunosorbent Assay (ELISA) Procedures

Blood obtaining procedures were modified from Mundermann et al. [3]. Participants were asked to limit their physical activity 48 hours prior to the experiment. On the day of the experiment, participants made their breakfast within one hour after waking up and the experiment started two to three hours after breakfast. In addition, participants were seated on a chair for 15-min immediately before the experiment. Five-milliliter blood samples were obtained by a certified research nurse from the same antecubital vein immediately before, immediately after, and 0.5 hours after a 30-min walking exercise. During the walking exercise of the test protocol, participants walked at a pace of 5 km/h on a treadmill with 1.5 % incline. After the walking exercise, participants sat on an office chair for 30-min and were asked to rest.

Blood sample collection and storage procedures were described previously [4]. Venous blood samples were obtained from vena mediana cubitii. After clotting for 60 min at room temperature, samples were centrifuged at 5000 rpm for 10-min. The serum samples were stored at -80°C until analysis.

Serum COMP concentrations were analyzed with a commercially available enzyme-linked immunosorbent assay based on two monoclonal antibodies: COMP ELISA and AnaMar Medical (Sweden). ELISA analysis was performed in a private institution and assay procedures were followed according to the manufacturer's guidelines. The order of blood samples was mixed and biochemist was blind to allocation of samples. All blood samples were analyzed simultaneously to maintain uniform specificity across individuals.

Statistical Procedures

The effects of 12 weeks interventions on general fitness and serum COMP concentrations at pre-tests and post-tests were analyzed using 4x2 (groups and time) mixed repeated measures ANOVA for each variable. Paired-samples t-tests were employed for comparison of the serum COMP concentrations during rest, fatigue and recovery states. In order to decrease the probability of committing type-1 error, a method of multiple comparisons by Bonferroni confidence interval adjustment was performed.

Sample size calculation was performed to eliminate type II error. Sample size was calculated using the G*Power 3.1.3 (Heinrich-Heine-University) software [5]. Significance level was set at 0.05 and a medium effect size (0.25) with two-sided calculation was used. Effect size contains the magnitude of difference between groups and values of 0.25, indicates medium effect of treatment [6]. By these assumptions, to achieve a power of 0.80, a sample size of 36 participants was necessary. Conservatively, 48 subjects were recruited since we expected a 20% dropout rate due to the demanding nature of the intervention program and our previous experience.

ELIGIBILITY:
Inclusion Criteria:

* body mass index lower than 30
* availability of participants for the tests and attendance to training sessions

Exclusion Criteria:

* osteoarthritis, rheumatoid arthritis or other inflammatory joint disease
* intra-articular steroid injection
* mal-alignment of the knees (varus/valgus) larger than 15°
* recent (within six months) fracture of lower extremity.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur Celik, PhD, Study Director — Middle East Technical University; Feza Korkusuz, PhD, Principal Investigator — Middle East Technical University
Locations (1):
- Middle East Technical University, Medical Center and Physical Education and Sports Dep., Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Mundermann A, Dyrby CO, Andriacchi TP, King KB. Serum concentration of cartilage oligomeric matrix protein (COMP) is sensitive to physiological cyclic loading in healthy adults. Osteoarthritis Cartilage. 2005 Jan;13(1):34-8. doi: 10.1016/j.joca.2004.09.007. PMID 15639635
- [Background] Andersson ML, Thorstensson CA, Roos EM, Petersson IF, Heinegard D, Saxne T. Serum levels of cartilage oligomeric matrix protein (COMP) increase temporarily after physical exercise in patients with knee osteoarthritis. BMC Musculoskelet Disord. 2006 Dec 7;7:98. doi: 10.1186/1471-2474-7-98. PMID 17156423
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Johnson EP. ACSM's Guidelines for Exercise Testing and Prescription. 6th ed. Baltimore: Lippincott, Williams and Wilkins, 2000.
- [Result] Bompa TO. Periodization : theory and methodology ot training. Champaign, IL: Human Kinetics, 1999.
- [Result] Field AP. Discovering Statistics Using SPSS for Windows: Advanced Techniques for Beginners. London: Sage Publications, Inc., 2000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Impact Loading | Moderate-Impact Loading | Non-Impact Loading | Control Group
Started | 12 | 12 | 12 | 12
Completed | 11 | 11 | 11 | 11
Not Completed | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Impact Loading | Moderate-Impact Loading | Non-Impact Loading | Control Group | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 11 | 11 | 44
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (1.3) | 21.1 (1.5) | 22.8 (1.9) | 22.6 (2.1) | 21.8 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 11 | 11 | 11 | 11 | 44
Region of Enrollment [Number; unit: participants]
  Turkey | 11 | 11 | 11 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum COMP Accumulation, Triggered by Acute Exercise, After 12 Weeks of Different Regular Exercises
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: U/l
Arm/Group | High-Impact Loading | Moderate-Impact Loading | Non-Impact Loading | Control Group
Number analyzed (Participants) | 11 | 11 | 11 | 11
U/l | -1.60 (0.95) | -0.53 (0.44) | -0.19 (1.70) | -0.12 (0.39)

2. Secondary Outcome: Physical (Body Mass Index) Changes of Participants
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Non-Impact Loading: Performed non-impact swimming exercise during intervention period.
- Control Group: Not participated any organized physical exercise
Arm/Group | High-Impact Loading | Moderate-Impact Loading | Non-Impact Loading | Control Group
Number analyzed (Participants) | 11 | 11 | 11 | 11
kg/m^2 | -0.73 (0.67) | -0.49 (0.54) | -0.72 (1.09) | -0.07 (0.65)

3. Secondary Outcome: Physiological (Maximum Oxygen Consumption) Changes of Participants
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- High-Impact Loading: Performed high-impact running exercise for 12 weeks
- Moderate-Impact Loading: Performed Moderate-impact cycling exercise for 12 weeks
- Non-Impact Loading: Performed Non-impact swimming exercise for 12 weeks
Arm/Group | High-Impact Loading | Moderate-Impact Loading | Non-Impact Loading | Control Group
Number analyzed (Participants) | 11 | 11 | 11 | 11
ml/kg/min | 4.91 (3.48) | 2.93 (2.20) | 5.46 (2.51) | 1.11 (3.32)

ADVERSE EVENTS:
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | High-Impact Loading | Moderate-Impact Loading | Non-Impact Loading | Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes